CLINICAL TRIAL: NCT01052441
Title: Iodine Content for Diagnostic AccuRacy and Patient Comfort For Individuals Undergoing Cardiac CT Scanning: The Multicenter ICARUS Trial
Brief Title: Iodine Content for Diagnostic AccuRacy and Patient Comfort For Individuals Undergoing Cardiac Computed Tomography (CT) Scanning
Acronym: ICARUS
Status: Completed | Type: Observational
Sponsor: MDDX LLC (Industry)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: GEH-CRLLC-1.2009
Record Dates: First submitted 2010-01-14; First posted 2010-01-20 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Coronary Arteriosclerosis
Keywords: CCTA; Coronary Artery Stenosis; Iodinated Contrast; Invasive Coronary Angiography
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CT Scan: Subjects with typical or atypical chest pain suspected of coronary artery disease and referred for an elective invasive coronary angiography (ICA), and scheduled to undergo CCTA before ICA or after ICA, if no intervention has been performed.

SUMMARY:
The purpose of the study is to evaluate diagnostic performance of high iodine (iopamidol 370 mg/dl) content versus low iodine (iodixanol 300 mg/dl) content for diagnostic accuracy by contrast-enhanced Coronary Cardiac Computed Tomography (CCTA) using a 64-detector-row CT scanner for detection of presence or absence of coronary artery obstruction when compared against invasive coronary angiography, the standard of truth.

DETAILED DESCRIPTION:
Coronary Cardiac CT (CCTA) is a widely accepted modality for non-invasive evaluation of coronary atherosclerosis. The diagnostic performance of CCTA for detecting coronary artery plaque burden has been validated in numerous studies, reaching a negative predictive value of 99%.

The current gold standard for anatomic coronary imaging is Invasive Coronary Angiography (ICA) which portends a small but significant procedural-related complication of 1.7%. Non-invasive coronary imaging has the potential to replace ICA but the variability in diagnostic performance of CCTA remains under study. Among the potential variables causing differences in diagnostic performance is perhaps the degree of opacification of coronary artery by iodinated contrast. While numerous contrast agents exist, those that provide improved low and high contrast resolution (for delineating plaque from arterial wall and lumen from plaque, respectively) are hypothetically, the most optimal agents. To date, however, this has not been well evaluated. Further, use of a contrast agent which maximizes patient comfort is desired, as this may reduce heart rate increases and heart rate variability, which may in turn improve diagnostic image quality of CCTA.

We hypothesize that the use of lower iodine content iso-osmolar agent - iodixanol - will improve diagnostic performance and patient comfort, as compared to higher iodine content low osmolar iodinated contrast - iopamidol.

ELIGIBILITY:
Inclusion Criteria:

* The subject is ≥18 years old.
* The subject has typical or atypical chest pain suspected of Coronary Artery Disease (CAD) and is referred for an elective coronary angiography.
* The subject must be scheduled to undergo a CATH procedure between 72 hours and 3 weeks of the CCTA procedure.
* The subject must not undergo any cardiac interventional treatment between the 2 procedures.
* The subject must have a sinus rhythm with stable heart rate of ≤75 beats per minute (bpm) and if heart rate is >65 bpm, the subject must agree to the use of beta-blocker(s) prior to the CT scan procedure to achieve stable heart rate of ≤65 bpm.

Exclusion Criteria:

* The subject has an established diagnosis of CAD by a) previous ICA, b) prior myocardial infarction confirmed by electrocardiogram (ECG), or c) prior revascularization (balloon angioplasty, stent placement, or coronary artery bypass grafting (CABG).
* The subject has a known allergy to iodinated contrast agent, including but not limited to hives, anaphylactoid or cardiovascular reactions, laryngeal edema and bronchospasm.
* The subject has impaired renal function with a serum creatinine level of 1.7 mg/dL (150 μmol/L) or above.
* The subject has atrial fibrillation/flutter or any irregular heart rhythm considered by the investigator to interfere with temporal acquisition of cardiac CT images.
* The subject has a resting heart rate of >100 bpm and/or a resting systolic blood pressure of <100 mm Hg.
* The subject has an artificial heart valve(s).
* The subject has had prior pacemaker or internal defibrillator lead implantation.
* The subject's resting heart rate is >65 bpm and beta-blocker therapy is contraindicated.
* The subject has a contraindication to Verapamil when beta-blocker therapy cannot be administered.
* The subject has a contraindication to nitroglycerin.
* The subject has evidence of ongoing or active clinical instability.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects are over 18 years or older. They have been referred to a cardiologist for suspected CAD and then scheduled for an elective invasive coronary angiography.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy for coronary artery stenosis detection at the per-segment, per-vessel and per-patient level using an 18-coronary artery segment model as defined by Society of Cardiovascular Computed Tomography (SCCT), as compared to ICA. | 72 hours

SECONDARY OUTCOMES:
Heart rate increase and variability during contrast injection. Rates of 7-day contrast-induced nephropathy. Any untoward adverse reactions like flushing, itching, nausea/vomiting etc | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Robert Benton, MD, Principal Investigator — Capital Cardiology Associates
Locations (3):
- United States (2):
  - Capital Cardiology Associates, Albany, New York
  - Hudson Valley Heart Center, Poughkeepsie, New York
- University of British Columbia, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Miller JM, Rochitte CE, Dewey M, Arbab-Zadeh A, Niinuma H, Gottlieb I, Paul N, Clouse ME, Shapiro EP, Hoe J, Lardo AC, Bush DE, de Roos A, Cox C, Brinker J, Lima JA. Diagnostic performance of coronary angiography by 64-row CT. N Engl J Med. 2008 Nov 27;359(22):2324-36. doi: 10.1056/NEJMoa0806576. PMID 19038879